CLINICAL TRIAL: NCT03275545
Title: Neural Correlates of Reward and Symptom Expression in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2017-25878
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anorexia Nervosa, Weight Restored: Individuals with a recent diagnosis of anorexia nervosa (within the past 6 months), who currently have their weight in a healthy range (BMI > or = 18.5 kg/m2)
  Interventions: Other: No intervention
- Non-eating disorder Control: Individuals without a history of an eating disorder and no current DSM-5 psychiatric diagnoses.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is being examined in this study

SUMMARY:
The objective of this study is to identify the patterns of brain activity in reward circuitry that promote symptoms of anorexia nervosa. This project will compare weight-restored individuals with anorexia nervosa to a non-eating disorder control group on reward brain circuitry patterns in response to typically rewarding cues (i.e., entertaining videos) and disorder-specific restrictive eating cues (i.e., low-fat food choice) using fMRI. In addition, this study will examine which neurobiological reward responses among weight-restored individuals with anorexia nervosa predict objective restrictive eating (measured by laboratory meal intake) and longitudinal risk of relapse one year later.

DETAILED DESCRIPTION:
Aim 1: To compare patterns of brain activity in reward circuits to typically rewarding cues and disorder-specific cues between weight-restored individuals with anorexia nervosa and non-eating disorder controls

Hypothesis 1a: Activity in reward circuitry will be elevated in response to typically rewarding cues in the non-eating disorder control group versus weight-restored anorexia nervosa group.

Hypothesis 1b: Activity in reward circuitry will be elevated in response to disorder-specific in the weight-restored anorexia nervosa group versus the non-eating disorder control group.

Aim 2: To specify the relationship between brain patterns related to reward and restrictive eating among weight-restored individuals with anorexia nervosa

Hypothesis 2a: Lower reward circuit activity in response to typically rewarding cues will predict lower test meal intake for weight-restored anorexia nervosa group versus the non-eating disorder control group.

Hypothesis 2b: Higher reward circuit activity in response to disorder-specific cues will predict lower test meal intake for the weight-restored anorexia nervosa group versus the non-eating disorder control group.

Aim 3: To identify the brain patterns in reward circuitry associated with the risk of relapse among weight-restored individuals with anorexia nervosa in the year following weight-restoration.

Hypothesis 3a: Lower reward circuit activity in response to typically rewarding cues will predict relapse in the weight-restored anorexia nervosa group.

Hypothesis 3b: Higher reward circuit activity in response to disorder-specific cues will predict relapse in the weight-restored anorexia nervosa group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Current BMI > 18.5 kg/m2
* Ability to read and speak in English
* Right-handed
* Weight restored Anorexia Nervosa group: 1) DSM-5 diagnosis of AN in the past 6 months, with the exception of body image disturbance and intense fear of weight gain criteria; 2) BMI < 18.5 kg/m2 within past 6 months

Exclusion Criteria:

* Medical instability or current pregnancy
* Current substance use disorder, psychosis, or bipolar-I disorder
* Contraindication for fMRI
* History of neurological disorder/injury (e.g., stroke; head injury with > 10 minutes loss of consciousness)
* Food allergy that cannot be accommodated through substitutions to the laboratory test meal
* Lacking capacity to consent
* Non-eating disorder Control group: Current DSM-5 Axis-I diagnosis or current or past eating disorder diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Many participants will be community individuals self-referred to participate through a flyer or other study advertisement. Individuals who are patients at The Emily Program eating disorder treatment facility who are in the process of weight-restoration or who have recently been weight-restored from anorexia nervosa may also be presented with a flyer by clinical staff at the program through the process outlined above. Participants will also be recruited from logs of individuals who had previously participated in studies in our lab and stated that they would like to be contacted for future studies and our active recruitment log.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Brain activation in reward circuits | Baseline
  Activation in regions of interest in reward brain circuitry (i.e., ventral tegmental area, nucleus accumbens) in response to typically-rewarding and disorder-specific tasks

SECONDARY OUTCOMES:
Restrictive eating | Baseline
  Caloric consumption from a laboratory test meal
Relapse | 12 months
  Relapse from anorexia nervosa, defined as: BMI < 18.5 kg/m2 and/or binge eating and/or purging > 1x/week for 3 consecutive months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haynos, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States